CLINICAL TRIAL: NCT06816823
Title: A Clinical Study of CAR-NK Cells (CL-NK-001) in Patients With Advanced Pancreatic Cancer
Brief Title: CAR-NK Cells (CL-NK-001) in Pancreatic Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhuan Liao, Prof., Changhai Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHEC2025-028
Record Dates: First submitted 2025-02-01; First posted 2025-02-10 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Pancreatic Cancer
Keywords: pancreatic cancer; CAR-NK
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CL-NK-001 (Experimental): Dose escalation of at least 3 dose levels
  Interventions: Biological: CL-NK-001

INTERVENTIONS:
Biological: CL-NK-001 — Dose level 1 (5 × 10^8 cells); dose level 2 (15 × 10^8 cells); dose level 3 (30 × 10^8 cells); additional dose levels (investigator's discretion).

SUMMARY:
This is a single-center, open-label, first-in-human, dose-escalation study in patients with pancreatic cancer.

DETAILED DESCRIPTION:
A dose-escalation study will evaluate the safety, tolerability and efficacy of CAR-NK cells (CL-NK-001) in patients with locally advanced, metastatic, or recurrent pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-70 years;
2. Locally advanced, metastatic, or recurrent pancreatic cancer, with immunohistochemical detection of eGR1 (membrane positive tumor cell rate >40% and expression intensity ≥2+), who have failed, been intolerant to or reject standard treatment;
3. At least 1 measurable lesion according to RECIST 1.1;
4. Have not received anti-tumor treatment for at least 4 weeks;
5. ECOG performance status of 0-2;
6. Estimated life expectancy more than 12 weeks;
7. Hematology: neutrophils ≥ 1.5×10^9/L, lymphocytes ≥ 0.8×10^9/L, hemoglobin ≥ 100 g/L, and platelets ≥ 75 × 10^9/L;
8. Blood biochemistry: total bilirubin ≤ 2×ULN, alanine aminotransferase ≤ 3×ULN, aspartate aminotransferase ≤ 3×ULN, and creatinine clearance ≥ LLN (Cockcroft-Gault formula);
9. Volunteer to participate in this clinical study and willing to sign written informed consent.

Exclusion Criteria:

1. Evidence of central nervous system involvement;
2. Have received adoptive cell therapy;
3. Patients with any uncontrolled active infection, including but not limited to: HBV, HCV, HIV, or treponema pallidum serology positive;
4. Vaccinated with a live attenuated vaccine within 3 months;
5. History of immunodeficiency;
6. Active autoimmune disease;
7. Have severe conditions, including but not limited to: (1) severe respiratory diseases; (2) severe cardiovascular diseases (previous history of CABG/PCI; myocardial infarction/unstable angina pectoris, congestive heart failure of NYHA III-IV, left ventricular ejection fraction < 50%, or poorly controlled hypertension within 6 months; QTc interval > 480ms, long or short QT syndrome; previous history of ventrical arrhythmia, or ventrical arrhythmia under anti-arrhythmic drugs/ICD); (3) poorly controlled diabetes and other metabolic diseases; (4) severe gastrointestinal diseases (severe gastrointestinal bleeding, severe diarrhea of CTCAE ≥ 2, or severe gastrointestinal obstruction needing intervention);
8. Possible severe adverse events, allergy or other contraindications to drugs or its component under study;
9. Pregnant or lactating women;
10. History of neurological or psychological disorders;
11. Not suitable to participate this clinical study judged by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | 42 days of first infusion
  Safety
Maximum tolerated dose (MTD) | 42 days of first infusion
  Tolerability
Treatment-emergent adverse event (TEAE) and treatment-emergent serious adverse event (TESAE) | 42 days of first infusion
  Safety
Number of participants with abnormal clinical laboratory parameters reported as TEAE | 42 days of first infusion
  Safety
Number of participants with abnormal vital signs reported as TEAE | 42 days of first infusion
  Safety
Number of participants with change from baseline in QT/QTc interval in electrocardiogram | 42 days of first infusion
  Safety

SECONDARY OUTCOMES:
Objective response rate (ORR) | 42 days of first infusion
  Efficacy
Disease control rate (DCR) | 42 days of first infusion
  Efficacy
Progression-free survival (PFS) | 6 months
  Efficacy
Overall survival (OS) | 6 months
  Efficacy
Patient-reported quality of life (QoL) | 42 days of first infusion
  Measured by the European Organization for Research and Treatment of Cancer quality-of-life questionnaire (EORTC QLQ-C30)
Patient-generated subjective global assessment (PG-SGA) | 42 days of first infusion
  Nutritional status measurement with a medical history section assessed by patients and a physical assessment section assessed by medical staff

CONTACTS AND LOCATIONS:
Overall Officials: Zhuan Liao, MD PhD, Principal Investigator — Changhai Hospital; Xuetao Cao, MD PhD, Principal Investigator — National Key Laboratory of Immunity & Inflammation
Locations (1):
- Changhai Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No